CLINICAL TRIAL: NCT05712993
Title: Comparative Study Between Transcoronoid and Infrazygomatic Anterior Maneuvers to Localize the Maxillary Nerve Under Ultrasound Guidance
Brief Title: Comparative Study Between Transcoronoid and Infrazygomatic Anterior Maneuvers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iraqi Board of medical specialties (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IraqBoard
Record Dates: First submitted 2023-01-16; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcoronoid (Experimental): participants are TN patients complain TN without secondary causes of trigeminal neuralgia underwent V2 targeting through coronoid notch
  Interventions: Procedure: V2 thermal radio frequency
- infrazygomatic anterior out of plane (Experimental): participants are TN patients complain TN without secondary causes of trigeminal neuralgia underwent V2 targeting through infrazygomatic anterior out of plane
  Interventions: Procedure: V2 thermal radio frequency

INTERVENTIONS:
Procedure: V2 thermal radio frequency — V2 targeted thermal radio frequency safely without sustained V3 stimulation

SUMMARY:
new technique in targeting V2 under ultrasound guidance

DETAILED DESCRIPTION:
the classical approach of V2 transcoronoin for practitioner is considered as difficult with significant failure rate with sustained V3 motor stimulation our approach infrazygomatic anterior out of plane is considered much easier in achieving pure V2 stimulation without V3 which make the thermal radio frequency 80 Celsius can be performed safely

ELIGIBILITY:
Inclusion Criteria:above 40 severe pain normal neurological examination -

Exclusion Criteria:metastasis allergy to medication used radio frequency precautions previous failed radio frequency or microvascular decompression gamma knife coagulpathy sepsis or active infection at site of needle entry

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
1-efficacy and safety of infrazygomatic anterior out of plane 2- how can infrazygomatic maneuver can help in decrease the chance of targeting V3 in addition V2 during injection | 2 years
  new method used to target V2 to decrease the chance of failure and to lessen the number of trials required the tools of measurement was the stimulation in volt and number of trial by No.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Mahdi, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
40 participants enrolled in the study complaining of sever TN with normal neurological examination